CLINICAL TRIAL: NCT03491800
Title: Patient and Family Partners in Heart Failure: Pilot Test of a Pre-visit Question Prompt List to Enhance Engagement of Heart Failure Patients and Family Members During Medical Visits
Brief Title: Patient and Family Partners in Heart Failure Care: Pilot Test of a Pre-visit Question Prompt List to Enhance Engagement During Medical Visits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); RTI International (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-2573; UL1TR001111 (NIH)
Record Dates: First submitted 2018-03-28; First posted 2018-04-09 (Actual); Results first posted 2020-08-13 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Individual patients and dyads (i.e., a HF patient and family member) will receive the question/topic prompt list immediately before their clinic visit
Masking Description: Given the nature of the intervention and it's intended purpose (i.e., to enhance communication with participants and health care providers), it is not possible to blind participants, care providers, or the investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Question/Topic Prompt List (Other): The Question/Topic Prompt List is provided to HF Patients and their family member (if applicable) for completion prior to being seen by the doctor.
  Interventions: Behavioral: Question/Topic Prompt List

INTERVENTIONS:
Behavioral: Question/Topic Prompt List — A written document containing suggested questions that the family member and/or patient may want to ask the health care provider during the visit. A section is included for the patient to check which behaviors they would like for their family member to engage in during the visit and space is provided for the family member to check which behaviors they are willing to perform during the visit.

SUMMARY:
The purpose of this study is to conduct a pilot study in 30 Heart Failure (HF) patients and visit companions (i.e., a family member who accompanies the patient to medical visits), to evaluate a pre- visit question/topic prompt list, designed to enhance patient and family member engagement during visits by providing a list of questions or topics that they may want to discuss with their health care provider.

DETAILED DESCRIPTION:
Participants in this study will include 30 HF patients or dyads (i.e., a patient and family member who accompanies the patient into the examination room at a visit). While our study primarily will target HF dyads, if the investigators encounter recruitment difficulties, unaccompanied HF patients (i.e., HF patients who do not have a family member who can participate in the study with them) will also be enrolled.

Procedures (methods): Single group pre-post study design.

After providing informed consent, HF patients or dyads will receive the prompt list while in the waiting room prior to their visit. Completing the prompt list involves two steps. In step 1, participants will independently select from a predetermined list of questions (within topic areas) that they would like to ask their health care provider. The questions/topics were developed by other HF patients and family members in another phase of the study. Also, patients will be asked to choose behaviors they would like their family member to engage in during the visit (e.g., write down the provider's instructions, ask questions), from a structured list developed based on prior research. Family members will identify which behaviors they are willing to perform. In step 2, patients or dyads will collectively prioritize which questions/topics to discuss during the visit. Each dyad member will receive a prompt list to complete in the clinic waiting room immediately before their appointment.

All visits will be audio-taped to assess effects of the intervention on communication behaviors during the visit. All participants will complete a questionnaire at baseline, 2 days after the audio-taped clinic visit, and at 3 months.

ELIGIBILITY:
Inclusion Criteria:

Patient Eligibility Criteria

* Ambulatory adult patients ≥ 30 years old
* Receive care in the University of North Carolina at Chapel Hill Cardiology practice
* Have a clinical diagnosis of HF
* Currently prescribed a loop diuretic
* Have a New York Heart Association class II-IV
* Must speak English
* Have a working telephone or live with the patient

Family Member Eligibility Criteria

* ≥ 18 years old and able to give informed consent
* Must be willing to participate in the intervention activities and provide informed consent
* Must speak English
* Have a working telephone or live with the patient

Health Care Provider Eligibility Criteria

* Must be an MD or advance practice provider (NP or PA) in the University of North Carolina at Chapel Hill Cardiology or General Internal Medicine practice
* Must be willing to have an enrolled patient visit audio-taped

Exclusion Criteria:

For patients:

* blindness,
* terminal illness with life expectancy <1 year (based on physician estimation),
* currently on or anticipated to start dialysis within 1 year,
* oxygen dependent chronic obstructive pulmonary disease,
* residency in a nursing home, or
* psychiatric illness that would interfere with protocol completion.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Wiley Cené, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC School of Medicine, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Accompanied Patients: The Question/Topic Prompt List is provided to Heart Failure (HF) Patients and their family member (if applicable) for completion prior to being seen by the doctor.
- Companions: Family members who accompanied enrolled patient participants to a visit and participated in the study with the patient.
- Unaccompanied Patients: The Question/Topic Prompt List is provided to individual, unaccompanied HF patient participants for completion prior to being seen by the doctor.
Period: Overall Study
Arm/Group | Accompanied Patients | Companions | Unaccompanied Patients
Started | 23 | 23 | 7
Completed | 23 | 23 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Accompanied Patients | Companions | Unaccompanied Patients | Total
Number analyzed (Participants) | 23 | 23 | 7 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (13.9) | 58.6 (16.0) | 61.1 (17.2) | 59.9 (3.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 19 | 5 | 30
  Male | 17 | 4 | 2 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 23 | 23 | 6 | 52
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 11 | 1 | 22
  White | 11 | 12 | 6 | 29
  More than one race | 2 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 23 | 7 | 53
Mean Score on the SCHFI - Maintenance Subscale [Mean (Standard Deviation); unit: units on a scale] — The Self-Care of Heart Failure Index (SCHFI) was used to measure self-care maintenance. The 10-item self-care maintenance scale assesses behaviors used to maintain physiologic stability (e.g., adherence to medications, frequent weighing).This subscale score is standardized, with scores ranging from 0-100 (higher scores indicates greater self-care confidence). Scores ≥ 70 are reflective of "adequate" self-care maintenance. A change in scale score of one-half of a standard deviation or more is considered clinically significant Population: This measure is completed by Accompanied and Unaccompanied Patients only. Data are missing for 1 Accompanied patient and 1 Unaccompanied patient and 23 Companions
  units on a scale
    number analyzed (Participants) | 22 | 0 | 6 | 28
    (all) | 76.20 (9.72) |  | 81.10 (12.76) | 77.25 (10.64)
Mean Score on the SCHFI - Management Subscale [Mean (Standard Deviation); unit: units on a scale] — The SCHFI was used to measure self-care management. The 10-item self-care management scale assesses decision-making in response to HF symptoms. The self-care management questions are answered and scored only if the respondent endorses having experienced dyspnea or ankle swelling within the past month. The subscale score is standardized, with scores ranging from 0-100 (higher scores indicates greater self-care management). Scores ≥ 70 are reflective of "adequate" self-care management. A change in scale score of one-half of a standard deviation or more is considered clinically significant. Population: This measure is completed by Accompanied and Unaccompanied patients only. Data are missing for 11 Accompanied patients and 3 Unaccompanied patients and all companions
  units on a scale
    number analyzed (Participants) | 12 | 0 | 4 | 16
    (all) | 69.17 (14.43) |  | 66.25 (6.29) | 68.44 (12.95)
Mean Score on the SCHFI - Confidence Subscale [Mean (Standard Deviation); unit: units on a scale] — The SCHFI 6-item subscale of the SCHFI assessed self-confidence in performing behaviors and making decisions to control heart failure symptoms. The subscale score is standardized with scores ranging from 0-100 (higher scores indicates greater self-care confidence). Scores ≥ 70 are reflective of "adequate" self-care confidence. A change in scale score of one-half of a standard deviation or more is considered clinically significant. Population: This measure is completed by Accompanied and Unaccompanied Patients only. Data are missing for 1 Accompanied patient and 1 Unaccompanied patient and all companions.
  units on a scale
    number analyzed (Participants) | 22 | 0 | 6 | 28
    (all) | 67.48 (19.44) |  | 60.23 (12.39) | 65.93 (18.40)
Mean Score on the CC-SCHFI - Maintenance Subscale [Mean (Standard Deviation); unit: units on a scale] — The Caregiver Contribution to Self-Care of Heart Failure Index (CC-SCHFI) is a 22-item measure (across 3 sub-scales) that assesses the contribution of caregivers to the self-care maintenance and self-care management of HF patients as well as their confidence in their ability to contribute to the patients' HF self-care. This 10- item subscale uses a 4-point Likert scale (never or rarely, sometimes, frequently, always or daily), with a standardized score from 0 to 100; higher scores indicate higher contribution to self-care maintenance. Population: This measure is completed by Companions only. Data are missing for 1 Companion and all accompanied and unaccompanied patients.
  units on a scale
    number analyzed (Participants) | 0 | 22 | 0 | 22
    (all) |  | 57.72 (23.37) |  | 57.72 (23.37)
Mean Score on the CC-SCHFI - Management Subscale [Mean (Standard Deviation); unit: units on a scale] — The CC-SCHFI is a 22-item measure (across 3 sub-scales) that assesses the contribution of caregivers to the self-care maintenance and self-care management of HF patients as well as their confidence in their ability to contribute to the patients' HF self-care. This 6-item subscale uses a 4-point Likert scale (never or rarely, sometimes, frequently, always or daily), with a standardized score from 0 to 100; higher scores indicate higher contribution to the patient's self-care management. Population: This measure is completed by Companions only. Data are missing for 1 Companion and all accompanied and unaccompanied patients.
  units on a scale
    number analyzed (Participants) | 0 | 22 | 0 | 22
    (all) |  | 75.56 (14.46) |  | 75.56 (14.46)
Mean Score on the CC-SCHFI - Confidence Subscale [Mean (Standard Deviation); unit: units on a scale] — The CC-SCHFI is a 22-item measure (across 3 sub-scales) that assesses the contribution of caregivers to the self-care maintenance and self-care management of HF patients as well as their confidence in their ability to contribute to the patients' HF self-care. This 6-item subscale uses a 4-point Likert scale (never or rarely, sometimes, frequently, always or daily), with a standardized score from 0 to 100; higher scores indicate higher confidence in their ability to contribute to the patient's self-care. Population: This measure is completed by Companions only. Data are missing for 1 Companion and all accompanied and unaccompanied patients.
  units on a scale
    number analyzed (Participants) | 0 | 22 | 0 | 22
    (all) |  | 68.24 (25.98) |  | 68.24 (25.98)
Mean Score on the PEPPI [Mean (Standard Deviation); unit: units on a scale] — The Perceived Efficacy in Patient-Physician Interactions (PEPPI) measure, a 6-item measure assessed confidence (self-efficacy) in communicating with health care providers. Each question is scored using a 5-point Likert scale (0 = not at all confident to 5 = very confident). Higher scores indicate greater confidence in communicating with health care providers. Population: Row total differs from overall total due to missing data on the questionnaire
  units on a scale
    number analyzed (Participants) | 22 | 22 | 7 | 51
    (all) | 3.68 (0.32) | 3.83 (0.31) | 3.52 (0.56) | 3.72 (0.38)
Mean Score on Communication With Physicians Measure [Mean (Standard Deviation); unit: units on a scale] — The Communication with Physicians measure is a 3-item measure which assesses the frequency of patients' engagement in communication behaviors during medical visits, including, preparing a list of questions, asking questions about treatment, and discussing personal problems with provider. Each question is answered using a 6-point Likert scale ranging from 0=never to 5=always. Higher scores indicate more active engagement in communication during medical visits. Population: The Communication with Physicians measure was not completed by companions. Data are missing for 1 Accompanied patient and 1 Unaccompanied patient
  units on a scale
    number analyzed (Participants) | 22 | 0 | 6 | 28
    (all) | 3.35 (1.31) |  | 3.00 (1.66) | 3.27 (1.40)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Eligible Participants Who Enroll
Description: The investigators will assess enrollment success into the study among those considered eligible. Investigators aim to have at least 50% of eligible participants enroll into the trial.
Time Frame: 6 months
Population: Includes all participants screened for enrollment into the study
Measure: Number; unit: percentage of participants
Groups:
- Patient and Companions: All patients and companions who were screened for eligibility and contacted by telephone for possible study participation
Arm/Group | Patient and Companions
Number analyzed (Participants) | 120
percentage of participants | 44

2. Secondary Outcome: Mean Acceptability Checklist Score
Description: The investigators will assess the perceived value of the checklist using a series of 11 questions developed for this study. Each question is scored using a 6-point Likert response scale where 1 = strongly disagree and 6 = strongly agree. Higher scores mean higher perceived value of the checklist.
Time Frame: Within 2 days after receiving checklist
Population: Data were reported when present and applicable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Accompanied Patients | Companions | Unaccompanied Patients
Number analyzed (Participants) | 23 | 23 | 7
score on a scale
  Easier to talk to doctor | 5.09 (1.16) | 5.04 (1.36) | 4.86 (1.46)
  Existing questions matched what I wanted to ask | 5.35 (1.30) | 5.13 (1.42) | 5.14 (0.69)
  Adequate time in waiting room to finish checklist | 5.48 (1.20) | 5.52 (1.20) | 5.29 (1.89)
  Easy to fill out: number analyzed (Participants) | 22 | 22 | 7
  Easy to fill out | 5.86 (0.35) | 5.95 (0.21) | 6.00 (0.00)
  Instructions clear and understandable: number analyzed (Participants) | 22 | 22 | 7
  Instructions clear and understandable | 5.95 (0.21) | 5.91 (0.29) | 5.29 (1.89)
  Easy to use during discussion with Dr: number analyzed (Participants) | 18 | 17 | 6
  Easy to use during discussion with Dr | 5.89 (0.32) | 5.94 (0.24) | 5.50 (1.23)
  Would use checklist at next appt: number analyzed (Participants) | 18 | 17 | 6
  Would use checklist at next appt | 5.00 (1.75) | 5.12 (1.58) | 4.33 (1.86)
  Checklist helped to get more questions asked: number analyzed (Participants) | 18 | 17 | 6
  Checklist helped to get more questions asked | 5.39 (1.34) | 5.35 (1.27) | 4.83 (1.60)
  Able to learn more from Dr using checklist: number analyzed (Participants) | 18 | 17 | 6
  Able to learn more from Dr using checklist | 5.28 (1.36) | 5.24 (1.39) | 4.50 (1.64)
  Clearer understanding of companion's concerns: number analyzed (Participants) | 20 | 17 | 0
  Clearer understanding of companion's concerns | 4.75 (1.94) | 5.53 (1.23) |
  Felt supported by companion due to checklist: number analyzed (Participants) | 20 | 0 | 0
  Felt supported by companion due to checklist | 5.25 (1.52) |  |

3. Secondary Outcome: Mean Score on the Self-Care of Heart Failure Index (SCHFI) - Management Subscale
Description: The SCHFI was used to measure self-care management. The 10-item self-care management scale assesses decision-making in response to HF symptoms. Of note, the self-care management questions are answered and scored only if the respondent endorses having experienced dyspnea or ankle swelling within the past month.The subscale score is standardized, with scores ranging from 0-100 (higher scores indicate greater self-care management). Scores ≥ 70 are reflective of "adequate" self-care management. A change in scale score of one-half of a standard deviation or more is considered clinically significant. Measured at Baseline and during the 1 Month Follow-Up.
Time Frame: Up to 1 month after clinic visit
Population: This measure is completed by Accompanied and Unaccompanied patients only. Companion responses are not applicable here and are captured in a separate outcome measure. Data are missing for 11 Accompanied patients and 3 Unaccompanied patients.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Accompanied Patients | Companions | Unaccompanied Patients
Number analyzed (Participants) | 12 | 0 | 4
score on a scale
  Baseline | 69.17 (14.43) |  | 66.25 (6.29)
  1 Month Follow-Up | 61.67 (31.72) |  | 62.50 (6.45)
Statistical Analysis 1: Comparison: Accompanied Patients; Test type: Superiority; p = 0.30, t-test, 2 sided; Mean Difference (Net) = 7.5, Standard Error of Mean 0.15

4. Secondary Outcome: Mean Score on the Self-Care of Heart Failure Index (SCHFI) - Maintenance Subscale
Description: The SCHFI was used to measure self-care maintenance. The 10-item self-care maintenance scale assesses behaviors used to maintain physiologic stability (e.g., adherence to medications, frequent weighing).This subscale score is standardized, with scores ranging from 0-100 (higher scores indicates greater self-care maintenance). Scores ≥ 70 are reflective of "adequate" self-care maintenance. A change in scale score of one-half of a standard deviation or more is considered clinically significant. Measured at Baseline and during the 1 Month Follow-Up.
Time Frame: Up to 1 month after clinic visit
Population: This measure is completed by Accompanied and Unaccompanied patients only. Companion responses are not applicable here and are captured in a separate outcome measure. Data are missing for 1 Accompanied patients and 1 Unaccompanied patients.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Accompanied Patients | Companions | Unaccompanied Patients
Number analyzed (Participants) | 22 | 0 | 6
score on a scale
  Baseline | 76.20 (9.72) |  | 81.10 (12.76)
  1 Month Follow-Up | 76.51 (12.70) |  | 76.66 (9.43)
Statistical Analysis 1: Comparison: Accompanied Patients; Test type: Superiority; p = 0.90, t-test, 2 sided; Mean Difference (Final Values) = -0.3, Standard Error of Mean 0.43
Statistical Analysis 2: Comparison: Unaccompanied Patients; Test type: Superiority; p = 0.30, t-test, 2 sided; Mean Difference (Final Values) = 4.44, Standard Error of Mean 0.26

5. Secondary Outcome: Mean Score Self-Care of Heart Failure Index (SCHFI) F-Up Month 1 - Confidence Subscale
Description: The 6-item subscale of the SCHFI was used to assess self-confidence in performing behaviors and making decisions to control heart failure symptoms. The subscale score is standardized, with scores ranging from 0-100 (higher scores indicates greater self-care confidence). Scores ≥ 70 are reflective of "adequate" self-care confidence. A change in scale score of one-half of a standard deviation or more is considered clinically significant. Measured at Baseline and during the 1 Month Follow-Up.
Time Frame: Up to 1 month after
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Accompanied Patients | Companions | Unaccompanied Patients
Number analyzed (Participants) | 22 | 0 | 6
score on a scale
  Baseline | 67.48 (19.44) |  | 60.23 (12.39)
  1 Month Follow-Up | 70.51 (15.67) |  | 61.16 (13.16)
Statistical Analysis 1: Comparison: Accompanied Patients; Test type: Superiority; p = 0.40, t-test, 2 sided; Mean Difference (Final Values) = -3.03, Standard Error of Mean -0.28
Statistical Analysis 2: Comparison: Unaccompanied Patients; Test type: Superiority; p = 0.85, t-test, 2 sided; Mean Difference (Final Values) = 0.93, Standard Error of Mean 0.22

6. Secondary Outcome: Mean Score on Caregiver Contribution to Self-Care of Heart Failure Index (CC-SCHFI) - Confidence Subscale
Description: The CC-SCHFI is a 22-item measure (across 3 sub-scales) that was used to assess the contribution of caregivers to the self-care maintenance and self-care management of HF patients as well as their confidence in their ability to contribute to the patients' HF self-care. This 6-item subscale uses a 4-point Likert scale (never or rarely, sometimes, frequently, always or daily), with a standardized score from 0 to 100; higher scores indicate higher confidence in ability to contribute to the patient's self-care. Measured at Baseline and during the 1 Month Follow-Up.
Time Frame: Up to 1 month after.
Population: This measure is completed by Companions only. Data are missing for 1 Companion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Accompanied Patients | Companions | Unaccompanied Patients
Number analyzed (Participants) | 0 | 22 | 0
score on a scale
  Baseline |  | 68.24 (25.98) |
  1 Month Follow-Up |  | 73.29 (22.02) |
Statistical Analysis 1: Comparison: Companions; Test type: Superiority; p = 0.21, t-test, 2 sided; Mean Difference (Final Values) = -5.05, Standard Error of Mean -0.25

7. Secondary Outcome: Mean Score on Caregiver Contribution to Self-Care of Heart Failure Index (CC-SCHFI) - Maintenance Subscale
Description: The CC-SCHFI is a 22-item measure (across 3 sub-scales) that assesses the contribution of caregivers to the self-care maintenance and self-care management of HF patients as well as their confidence in their ability to contribute to the patients' HF self-care. This 10- item subscale uses a 4-point Likert scale (never or rarely, sometimes, frequently, always or daily), with a standardized score from 0 to 100; higher scores indicate higher contribution to self-care maintenance. Measured at Baseline and during the 1 Month Follow-Up.
Time Frame: Up to 1 month after
Population: This measure is completed by Companions only. Patient responses are not applicable here and are captured in a separate outcome measure. Data are missing for 1 Companion.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Accompanied Patients | Companions | Unaccompanied Patients
Number analyzed (Participants) | 0 | 22 | 0
score on a scale
  Baseline |  | 57.72 (23.37) |
  1 Month Follow-Up |  | 57.42 (26.18) |
Statistical Analysis 1: Comparison: Companions; Test type: Superiority; p = 0.95, t-test, 2 sided; Mean Difference (Final Values) = 0.30, Standard Error of Mean 0.23

8. Secondary Outcome: Mean Score on Caregiver Contribution to Self-Care of Heart Failure Index (CC-SCHFI) - Management Subscale
Description: The CC-SCHFI is a 22-item measure (across 3 sub-scales) that assesses the contribution of caregivers to the self-care maintenance and self-care management of HF patients as well as their confidence in their ability to contribute to the patients' HF self-care. This 6-item subscale uses a 4-point Likert scale (never or rarely, sometimes, frequently, always or daily), with a standardized score from 0 to 100; higher scores indicate higher contribution to the patient's self-care management. Measured at Baseline and during the 1 Month Follow-Up.
Time Frame: Up to 1 month after
Population: This measure is completed by Companions only. Accompanied and Unaccompanied responses are not applicable here and are captured in a separate outcome measure. Data are missing for 14 Companions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Accompanied Patients | Companions | Unaccompanied Patients
Number analyzed (Participants) | 0 | 9 | 0
score on a scale
  Baseline |  | 75.56 (14.46) |
  1 Month Follow-Up |  | 72.22 (14.81) |
Statistical Analysis 1: Comparison: Companions; Test type: Superiority; p = 0.52, t-test, 2 sided; Mean Difference (Final Values) = 3.34, Standard Error of Mean -0.20

9. Secondary Outcome: Mean Score on Perceived Efficacy in Patient-Physician Interactions (PEPPI)
Description: The PEPPI is a 6-item measure which assesses confidence (self-efficacy) in communicating with health care providers. Each question is scored using a 5-point likert scale (0= not at all confident to 5=very confident). Higher scores indicate greater confidence in communicating with health care providers. Measured at Baseline, 2-Day Follow-Up, and during the 1 Month Follow-Up.
Time Frame: Up to 1 month after clinic visit
Population: Reported data are less than the total number of participants who completed each arm due to participants not responding to questions for this measure. Data are missing for 1 Accompanied, 1 Unaccompanied, and 1 Companion.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Accompanied Patients | Companions | Unaccompanied Patients
Number analyzed (Participants) | 22 | 22 | 6
score on a scale
  Baseline | 3.68 (0.32) | 3.83 (0.31) | 3.52 (0.56)
  1 Month Follow-Up | 3.76 (0.29) | 3.81 (0.33) | 3.78 (0.39)
Statistical Analysis 1: Comparison: Accompanied Patients; Test type: Superiority; p = 0.23, t-test, 2 sided; Mean Difference (Final Values) = -38.25, Standard Error of Mean -38.25
Statistical Analysis 2: Comparison: Companions; Test type: Superiority; p = 0.67, t-test, 2 sided; Mean Difference (Final Values) = 0.02, Standard Error of Mean 22
Statistical Analysis 3: Comparison: Unaccompanied Patients; Test type: Superiority; p = 0.054, t-test, 2 sided; Mean Difference (Final Values) = -0.26, Standard Error of Mean 9.62

10. Secondary Outcome: Mean Score on Communication With Physicians Measure
Description: The Communication with Physicians measure by Lorig was used. It is a 3-item measure assessing the frequency of patients' engagement in communication behaviors during medical visits, including, preparing a list of questions, asking questions about treatment, and discussing personal problems with provider. Each question is answered using a 6-point Likert scale ranging from 0=never to 5=always. Higher scores indicate more active engagement in communication during medical visits. Measured at Baseline and during the 1 Month Follow-Up.
Time Frame: Up to 1 month after clinic visit
Population: This measure was only answered by patients. Companion responses are not applicable here. Data are missing for 1 Accompanied patients and 1 Unaccompanied patients.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Accompanied Patients | Companions | Unaccompanied Patients
Number analyzed (Participants) | 22 | 0 | 6
score on a scale
  Baseline | 3.35 (1.31) |  | 3.00 (1.66)
  1 Month Follow-Up | 3.45 (0.99) |  | 2.72 (0.98)
Statistical Analysis 1: Comparison: Accompanied Patients; Test type: Superiority; p = 0.60, t-test, 2 sided; Mean Difference (Final Values) = -0.1, Standard Error of Mean 5.4
Statistical Analysis 2: Comparison: Unaccompanied Patients; Test type: Superiority; p = 0.40, t-test, 2 sided; Mean Difference (Final Values) = 0.28, Standard Error of Mean 3.29

ADVERSE EVENTS:
Time Frame: Not applicable as safety data were not collected during the study
Description: Safety data were not planned to be collected during the study.
Arm/Group | Accompanied Patients | Companions | Unaccompanied Patients
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT03491800/Prot_SAP_000.pdf